CLINICAL TRIAL: NCT01513317
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multicenter Study Comparing Siltuximab Plus Best Supportive Care to Placebo Plus Best Supportive Care in Anemic Subjects With International Prognostic Scoring System Low- or Intermediate-1-Risk Myelodysplastic Syndrome
Brief Title: A Study Comparing Siltuximab Plus Best Supportive Care to Placebo Plus Best Supportive Care in Anemic Patients With International Prognostic Scoring System Low- or Intermediate-1-Risk Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped after the interim analysis based on lack of sufficient efficacy. There were no safety concerns.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR100752; CNTO328MDS2001 (Other: Janssen Research & Development, LLC); 2011-000261-12 (EudraCT Number)
Record Dates: First submitted 2011-10-21; First posted 2012-01-20 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; MDS; Blood and lymphatic diseases; Siltuximab; Anemic
MeSH Terms: conditions — Myelodysplastic Syndromes; Lymphatic Diseases | interventions — siltuximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Siltuximab (Experimental): 15 mg/kg of siltuximab administered as a 1-hour infusion every 4 weeks + best supportive care (BSC)
  Interventions: Drug: Siltuximab; Drug: Best supportive care (BSC)
- Placebo (Experimental): Placebo administered as a 1-hour infusion every 4 weeks + BSC
  Interventions: Drug: Placebo; Drug: Best supportive care (BSC)

INTERVENTIONS:
Drug: Siltuximab — 15 mg/kg administered as a 1-hour intravenous infusion every 4 weeks
  Arms: Siltuximab
Drug: Placebo — Administered as a 1-hour intravenous infusion every 4 weeks
  Arms: Placebo
Drug: Best supportive care (BSC) — Best supportive care according to local standards and guidelines

SUMMARY:
The purpose of this study is to evaluate the efficacy of siltuximab, demonstrated by a reduction in red blood cell (RBC), transfusions to treat the anemia of Myelodysplastic Syndrome (MDS).

DETAILED DESCRIPTION:
The study treatments will be administered double-blind for 12 weeks, meaning that the patient and study personnel will not know the identity of the treatment. Approximately 75 patients will be randomized (patients are assigned to a treatment by a chance) in a 2:1 ratio to receive siltuximab plus best supportive care (BSC) (Group A) or placebo plus BSC (Group B). BSC includes RBC transfusion, antimicrobials, white blood cell (WBC) growth factors, and platelet transfusions. Patients who complete 12 weeks of treatment may qualify to receive siltuximab as open-label (identity of treatment will be known) treatment. Treatment may continue until death, unacceptable toxicity, withdrawal of consent, or the clinical cutoff (defined as 24 weeks after the last patient is randomized), whichever occurs first. The study will end approximately 36 weeks after the last patient is randomized. Patient safety will be monitored. Siltuximab and matching placebo will be supplied as a sterile, lyophilized formulation for reconstitution and intravenous (IV) infusion. Group A: siltuximab (15 mg/kg) administered as a 1-hour infusion every 4 weeks + BSC, or Group B: placebo administered as a 1-hour infusion every 4 weeks + BSC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of myelodysplastic syndrome (MDS), according to World Heath Organization or the French-American-British Cooperative Group pathologic classification, with an International Prognostic Scoring System score 0, 0.5, or 1.0, indicating Low- or INT-1-risk disease.
* Documented RBC transfusion of at least 2 units of RBC for the treatment of the anemia of MDS in the 8 weeks preceding the start of the Screening Period.
* Adequate iron stores, demonstrated by either the presence of stainable iron in the bone marrow or a serum ferritin of > 100 ng/mL.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2.
* Symptomatic anemia (defined by a score > 0 on the Non-Chemotherapy Anemia Symptom Scale [NCA-SS]).

Exclusion Criteria:

* Had treatment with drugs or other agents targeting IL-6 or its receptor within 4 weeks of randomization.
* Any condition that, in the opinion of the investigator, would make participation not in the best interest (eg, compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments.
* Patients with Chronic Myelomonocytic Leukemia (CMML).
* Causes other than MDS contributing to anemia, such as Vitamin B12 or folate deficiency, bleeding, hemolysis, hemoglobinopathy, or chronic renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (23):
- United States (5):
  - Tampa, Florida
  - Boston, Massachusetts
  - New York, New York
  - Winston-Salem, North Carolina
  - Houston, Texas
- Australia (3):
  - Box Hill
  - Camperdown
  - St Leonards
- Belgium (4):
  - Antwerp
  - Bruges
  - Ghent
  - Yvoir
- Netherlands (2):
  - Dordrecht
  - The Hague
- Russia (3):
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
- Spain (5):
  - Barcelona
  - Madrid
  - Oviedo (Asturias)
  - Salamanca
  - Valencia
- Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 76 participants were enrolled at 6 sites in Spain, 5 sites in the United States, 4 sites in Belgium, 3 sites each in Australia and the Russian Federation, 2 sites in the Netherlands, and 1 site in Sweden.
Pre-assignment Details: All 76 participants were enrolled and randomly assigned in the study.
Groups:
- Placebo: Placebo administered as a 1-hour infusion every 4 weeks + best supportive care (BSC)
Period: Overall Study
Arm/Group | Siltuximab | Placebo
Started | 50 | 26
Completed | 16 | 2
Not Completed | 34 | 24
Not completed — Withdrawal by Subject | 15 | 4
Not completed — Death | 1 | 1
Not completed — Study terminated by sponsor | 18 | 18
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Siltuximab | Placebo | Total
Number analyzed (Participants) | 50 | 26 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (7.7) | 72 (7.61) | 70.8 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 9 | 32
  Male | 27 | 17 | 44
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 2 | 5
  Belgium | 4 | 4 | 8
  Netherlands | 2 | 1 | 3
  Russian Federation | 5 | 3 | 8
  Spain | 10 | 5 | 15
  Sweden | 3 | 0 | 3
  United States | 23 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Reduction in Red Blood Cell (RBC) Transfusions to Treat Anemia of Myelodysplastic Syndrome (MDS)
Description: Reduction in RBC transfusions to treat the anemia of MDS is defined as a ≥50 percentage relative decrease and a ≥2 unit absolute decrease in RBC transfusions in the 8 weeks before the unblinding (scheduled to occur after 12 weeks of treatment) compared with RBC transfusions in the 8 weeks before the date the informed consent form was signed.
Time Frame: Up to Week 13
Population: Intent-to-treat population: Included all randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 50 | 26
Percentage of participants | 12 | 3.8
Statistical Analysis 1: Comparison: Siltuximab vs Placebo; Test type: Superiority or Other; p = 0.271, Cochran-Mantel-Haenszel; Difference in proportions = 0.082, 95% CI 2-sided [-0.03 to 0.20] — The estimated parameter is the difference in proportion of participants who had a reduction in RBC transfusion to treat the anemia of MDS

2. Secondary Outcome: Change From Baseline in the Mean Hemoglobin Concentrations at Week 13
Time Frame: Baseline and Week 13
Population: Intent-to-treat population: Included all randomized participants with evaluable data at Week 13
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 31 | 18
g/dL | -0.07 (1.503) | -0.13 (1.375)
Statistical Analysis 1: Comparison: Siltuximab vs Placebo; Test type: Superiority or Other; p = 0.872, ANCOVA; Difference in LS means = 0.07, 95% CI 2-sided [-0.79 to 0.93] — The estimated parameter is the difference in LS means of the change from baseline hemoglobin levels at Week 13

3. Secondary Outcome: Percentage of Participants Achieving Hemoglobin Improvement (≥1.5 g/dL Increase From Baseline) Unrelated to Red Blood Cell (RBC) Transfusion at Week 13
Time Frame: Week 13
Population: Intent-to-treat population: Included all randomized participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 50 | 26
Percentage of Participants | 8.0 | 3.8
Statistical Analysis 1: Comparison: Siltuximab vs Placebo; Test type: Superiority or Other; p = 0.494, Cochran-Mantel-Haenszel; Difference in proportions = 0.042, 95% CI 2-sided [-0.06 to 0.15] — The estimated parameter is the difference in proportion of participants achieving hemoglobin improvement at Week 13

4. Secondary Outcome: Percentage of Participants Who Did Not Require a Red Blood Cell (RBC) Transfusions to Treat Anemia of Myelodysplastic Syndrome (MDS) in the 8 Weeks of Treatment Before Unblinding at Week 13
Time Frame: 8 weeks
Population: Intent-to-treat population: Included all randomized participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 50 | 26
Percentage of Participants | 4.0 | 3.8
Statistical Analysis 1: Comparison: Siltuximab vs Placebo; Test type: Superiority or Other; p = 0.986, Cochran-Mantel-Haenszel; Difference in proportions = 0.002, 95% CI 2-sided [-0.09 to 0.09] — The estimated parameter is the difference in proportion of participants who did not require a blood transfusion in the 8 weeks of treatment before unblinding at Week 13

5. Secondary Outcome: Mean Changes From Baseline in Percentages of Bone Marrow Blast Cells at Week 13
Time Frame: Baseline and Week 13
Population: Intent-to-treat population: Included all randomized participants with evaluable data at Week 13
Measure: Mean (Standard Deviation); unit: Percentage of Bone Marrow Blast Cells
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 31 | 15
Percentage of Bone Marrow Blast Cells | 2.1 (8.22) | 0.2 (2.08)
Statistical Analysis 1: Comparison: Siltuximab vs Placebo; Test type: Superiority or Other; p = 0.363, ANCOVA; Difference in LS means = 1.96, 95% CI 2-sided [-2.35 to 6.27] — The estimated parameter is the difference in LS means for changes from baseline in bone marrow blasts at Week 13

6. Secondary Outcome: Median Number of Red Blood Cell (RBC) Transfusions to Treat Anemia of Myelodysplastic Syndrome (MDS) During the 8 Weeks of Treatment Before Unblinding at Week 13
Time Frame: 8 weeks
Population: Intent-to-treat population: Included all randomized participants who completed Week 13 unblinding
Measure: Median (Full Range); unit: RBC Transfusions
Arm/Group | Siltuximab | Placebo
Number analyzed (Participants) | 36 | 22
RBC Transfusions | 6.0 [0 to 14] | 6.5 [0 to 25]
Statistical Analysis 1: Comparison: Siltuximab vs Placebo; Test type: Superiority or Other; p = 0.073, ANCOVA; Difference in LS means = -1.69, 95% CI 2-sided [-3.55 to 0.17] — The estimated parameter is the difference in LS means of the number of RBC transfusions during the 8 weeks of treament before unblinding at Week 13

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the time period between the first dose of study medication through 30 days after the last dose.
Description: Safety was analyzed for all randomized participants who received at least 1 dose of study medication.
Arm/Group | Siltuximab | Placebo
Serious Adverse Events (participants affected / at risk) | 10/50 | 8/26
Other Adverse Events (participants affected / at risk) | 30/50 | 18/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab (N=50) | Placebo (N=26)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Cardiovascular Insufficiency (Cardiac disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Femoral Hernia (Gastrointestinal disorders) | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Mucosal Haemorrhage (General disorders) | 0 | 1
Cirrhosis Alcoholic (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Escherichia Bacteraemia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab (N=50) | Placebo (N=26)
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 2 | 2
Oedema Peripheral (General disorders) | 8 | 2
Hepatic Function Abnormal (Hepatobiliary disorders) | 5 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Hypotension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days